CLINICAL TRIAL: NCT04190095
Title: Developing Real-time Interaction and Motion Tracking in Immersive VR for Telerehabilitation
Brief Title: Real-time Interaction and Motion Tracking in VR for Telerehabilitation
Acronym: MoVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Wyoming (Other)
Responsible Party: Principal Investigator, Qin Zhu, Associate Professor, University of Wyoming
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 201901004QZ02535
Record Dates: First submitted 2019-12-03; First posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- User Interaction with Device (Experimental): A user will wear motion sensors and VR device to interact with object or another user in VR environment
  Interventions: Device: Motion Tracking in VR; Behavioral: VR Interaction

INTERVENTIONS:
Device: Motion Tracking in VR — Participant will wear motion sensors and VR devices
Behavioral: VR Interaction — Participant will perform VR interaction task

SUMMARY:
Current technology for telerehabilitation is limited to be audio- or video- based interaction without an objective and accurate measure of motor functions. A technology integrating motion tracking with 3D immersive virtual reality has been developed by an interdisciplinary team to shift the paradigm of telerehabilitation. We aim to take the significant step to develop the patient-centered telerehabilitation that will feature real-time patient-therapist interaction with functions of tele-monitoring, tele-diagnosis, and tele-therapy. Such an interactive telerehabilitation is expected to increase patient adherence to therapy and minimize the existing health disparities.

DETAILED DESCRIPTION:
By innovatively integrating the 3D motion tracking with 3D immersive virtual reality (VR), the real-time user interaction and simultaneous motion tracking and analysis in the immersive VR environment were made possible. We now propose to customize this technology for telerehabilitation. The ultimate goal is to build a VR-based interactive tele-rehab system that is patient-centered, with augmented feedback and tele-presence of therapist to assist rehabilitative exercises and recovery of motor functions in both real and virtual environment. To achieve this goal, we are specifically tackling three problems.

* 1: Cross validating the precision of motion data captured in VR. We will modify our current software (Unity-based) so that it can work simultaneous with two motion tracking systems (Optical tracking and Magnetic tracking) to capture motion data in a 3D VR environment. The recorded data in our software will be compared and correlated with those data recorded by the two motion tracking systems in 3D for examination of accuracy.
* 2: Building and testing the network code for remote data transmission and interaction. We will write network code to enable the remote transmission of motion tracking data between two sites. The latency of data transmission will be tested to determine the minimum speed of internet for implementing such a tele-rehab system.
* 3: Designing and implementing a VR interaction task for remote monitoring and diagnosis. A 3D interactive VR task will be built for real-time local interaction and the remote monitoring, assessment and intervention.

ELIGIBILITY:
Inclusion Criteria:

* Only the key researchers of this project can participate in the study

Exclusion Criteria:

* Any individual who is not the responsible researcher in this project shall not participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Tracking Accuracy | through study completion, approximately 1 year
  matching the motion trajectories in VR and REAL with a small error indicating a good match
Latency of Data Transmission | through study completion, approximately 1 year
  The duration for the tracked motion data to be transmitted to a remote computer
Total number of the basketed apples | through study completion, approximately 1 year
  Computer display of the total count of successfully picked and basketed apples from the tree

SECONDARY OUTCOMES:
Total excursion of the hand | through study completion, approximately 1 year
  The total distance (in CM) that the hand has traveled in space while performing the apple picking task
Mean speed of hand movement | through study completion, approximately 1 year
  The total excursion of the hand divided by 60 seconds (cm/s)

IPD SHARING:
Plan to Share IPD: No